CLINICAL TRIAL: NCT00531934
Title: A Randomized, Open Label Study to Evaluate the Effect of Doxycycline on Tarceva-induced Skin Rash in Patients With Non-small Cell Lung Cancer After Failure of First Line Chemotherapy
Brief Title: A Study of Management of Tarceva - Induced Rash in Patients With Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20829
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Doxycline; Drug: erlotinib [Tarceva]
- 2 (Active Comparator)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: Doxycline — 100mg po daily
  Arms: 1
Drug: erlotinib [Tarceva] — 150mg po daily

SUMMARY:
This 2 arm study will evaluate the management of Tarceva-induced skin rash in patients with non-small cell lung cancer who have failed first-line chemotherapy for advanced disease. Eligible patients will be randomized to receive a)doxycycline 100mg po daily or b)no preventative treatment; all patients will receive Tarceva 150mg/kg po daily. The anticipated time on study treatment is until disease progression or intolerable toxicity, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* confirmed non-small cell lung cancer;
* failure after first line chemotherapy for advanced disease, and scheduled for second line therapy with Tarceva.

Exclusion Criteria:

* rash of any etiology at study entry;
* history of significant heart disease;
* any other malignancies (other than adequately treated squamous cell skin cancer, or in situ cancer of the cervix);
* history of allergic reactions to tetracyclines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- France (21):
  - Antibes
  - Bordeaux
  - Brest
  - Caen
  - Chalon-sur-Saône
  - Chartres
  - Draguignan
  - Gap
  - Gleizé
  - Limoges
  - Metz
  - Nîmes
  - Paris
  - Perpignan
  - Périgueux
  - Pierre-Bénite
  - Pontoise
  - Rennes
  - Rouen
  - Tours
  - Vannes

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib Plus (+) Doxycycline: Participants received erlotinib 150 milligrams per day (mg/day), tablets, orally (PO) until progression or unacceptable toxicity and doxycycline 100 mg/day, tablets, PO for the first 4 months of the study; after this period it was the investigator's choice to continue treatment with doxycycline.
- Erlotinib: Participants received erlotinib 150 mg/day, tablets, PO until progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Erlotinib Plus (+) Doxycycline | Erlotinib
Started | 73 | 74
Completed | 7 | 11
Not Completed | 66 | 63
Not completed — Adverse Event | 4 | 8
Not completed — Progression | 52 | 42
Not completed — Death | 7 | 10
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population (ITT): all randomized participants who received at least
  1 dose of erlotinib.
Groups:
- Erlotinib + Doxycycline: Participants received erlotinib 150 mg/day, tablets, PO until progression or unacceptable toxicity and doxycycline 100 mg/day, tablets, PO for the first 4 months of the study; after this period it was the investigator's choice to continue treatment with doxycycline.
- Total: Total of all reporting groups
Arm/Group | Erlotinib + Doxycycline | Erlotinib | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.6) | 64.2 (11.1) | 63.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 48 | 50 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Skin Rash (Folliculitis) of Any Grade During the First 4 Months of Treatment
Description: Description of skin rash (folliculitis, including erythema, papulo-pustules, nodule, and crust) was according to Common Terminology Criteria for Adverse Events (CTCAE) version 3 scale. Medical pictures of the face (front and sides views) systematically, and of any region presenting with skin lesions were obtained. The pictures were reviewed by a centralized committee of evaluation.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population; data for 1 participant in the erlotinib treatment group were missing.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 73
percentage of participants | 71.2 | 80.8
Statistical Analysis 1: Comparison: Erlotinib + Doxycycline vs Erlotinib; Test type: Superiority or Other; p = 0.175, Chi-squared

2. Secondary Outcome: Number of Skin Rash (Folliculitis) Events During the First 4 Months of Treatment
Description: A cutaneous rash as folliculitis can be defined with several types including erythema, papulo-pustular and nodules.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: rash events
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
rash events | 57 | 62

3. Secondary Outcome: Percentage of Participants With Skin Rash (Folliculitis) During the First 4 Months of Treatment By Type
Description: A cutaneous rash as folliculitis can be defined with several types including erythema, papulo-pustule, nodule, and crust.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants
  Erythema | 55.8 | 70.7
  Papulo-pustule | 65.4 | 72.4
  Nodule | 1.9 | 0
  Crust | 9.6 | 25.9

4. Secondary Outcome: Percentage of Participants With Skin Rash (Folliculitis) During the First 4 Months of Treatment By Maximal Intensity
Description: Intensity of skin rashes was classified according to CTCAE grading. Grade 1 equals (=) Macular or papular eruption or erythema without associated symptoms; Grade 2=Macular or papular eruption or erythema with pruritus or other associated symptoms; localized desquamation or other lesions covering less than (<)50 percent (%) of body surface area (BSA); Grade 3=Severe, generalized erythroderma or macular, papular, or vesicular eruption; desquamation.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population; only participants with an adverse event of skin rash (folliculitis) during the first 4 months were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 52 | 59
percentage of participants
  Grade 1 | 61.5 | 18.6
  Grade 2 | 34.6 | 62.7
  Grade 3 | 3.8 | 18.6
Statistical Analysis 1: Comparison: Erlotinib + Doxycycline vs Erlotinib; Erlotinib + doxycycline vs Erlotinib: Grade 3 intensity skin rash (folliculitis); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants With at Least One Skin Rash (Folliculitis) of Any Grade After the First 4 Months of Treatment
Time Frame: Months 7, 10, and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 2.7 | 1.4

6. Secondary Outcome: Number of Skin Rash (Folliculitis) Events After the First 4 Months of Treatment
Description: A cutaneous rash as folliculitis can be defined with several types including erythema, papulo-pustular and nodules.
Time Frame: Months 7, 10, and 12
Population: ITT population
Measure: Number; unit: rash events
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 73
rash events | 2 | 1

7. Secondary Outcome: Number of Participants With Skin Rash (Folliculitis) After the First 4 Months of Treatment By Type
Description: as for outcome 3
Time Frame: Months 7, 10, and 12
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
participants
  Erythema | 1 | 1
  Papulo-pustule | 1 | 1
  Nodule | 0 | 0
  Crust | 0 | 0

8. Secondary Outcome: Number of Participants With Skin Rash (Folliculitis) After the First 4 Months of Treatment By Intensity
Description: Intensity of skin rashes was classified according to CTCAE grading. Grade 1=Macular or papular eruption or erythema without associated symptoms; Grade 2=Macular or papular eruption or erythema with pruritus or other associated symptoms; localized desquamation or other lesions covering <50% of BSA; Grade 3=Severe, generalized erythroderma or macular, papular, or vesicular eruption; desquamation.
Time Frame: Months 7, 10, and 12
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
participants
  Initial intensity: Grade 1 | 2 | 1
  Maximal intensity: Grade 1 | 2 | 1

9. Secondary Outcome: Time Free From Skin Rash (Folliculitis) During the First 4 Months of Treatment - Number of Participants With an Event
Description: Period without occurrence was determined as the number of days from the first dose of medication until the first appearance of folliculitis, analyzed using Kaplan-Meier analysis.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
participants | 52 | 59

10. Secondary Outcome: Time Free From Skin Rash (Folliculitis) During the First 4 Months of Treatment - Time to Event
Description: as for outcome 9
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
days | 14 [13 to 22] | 13 [8 to 16]
Statistical Analysis 1: Comparison: Erlotinib + Doxycycline vs Erlotinib; Test type: Superiority or Other; p = 0.143, Log Rank; Hazard Ratio (HR) = 0.763, 95% CI 2-sided [0.525 to 1.109]

11. Secondary Outcome: Percentage of Participants Estimated to be Event Free at 4 Months
Description: Percentage of participants estimated to be without skin rash (folliculitis) at 4 months.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 24.7 | 11.2

12. Secondary Outcome: Time Free From Skin Rash (Folliculitis) During the Whole Treatment Period - Number of Participants With an Event
Description: as for outcome 9
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 73
participants | 53 | 59

13. Secondary Outcome: Time Free From Skin Rash (Folliculitis) During the Whole Treatment Period - Time to Event
Description: as for outcome 9
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 73
days | 14 [13 to 22] | 13 [8 to 16]
Statistical Analysis 1: Comparison: Erlotinib + Doxycycline vs Erlotinib; Test type: Superiority or Other; p = 0.153, Log Rank; Hazard Ratio (HR) = 0.769, 95% CI 2-sided [0.529 to 1.116]

14. Secondary Outcome: Percentage of Participants Estimated to be Event Free at 12 Months
Description: Percentage of participants estimated to be without skin rash (folliculitis) at 12 months.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 19.8 | 11.2

15. Secondary Outcome: Duration of Skin Rash (Folliculitis) During the First 4 Months of Treatment
Description: If the cutaneous rash was ongoing at the last visit or Month 4, the duration of cutaneous rash was calculated between start of folliculitis and Visit Month 4 or premature withdrawal visit or death.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT Population; only participants with an event (folliculitis) were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 57 | 61
days | 59.6 (35.9) | 60.6 (33.5)

16. Secondary Outcome: Duration of Skin Rash (Folliculitis) During the Whole Treatment Period
Description: If the end of cutaneous rash was missing, the duration of cutaneous rash was calculated between start of folliculitis and last evaluation date.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population; only participants with an event (folliculitis) were included in the analysis.
Measure: Median (Standard Deviation); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 59 | 62
days | 86.7 (81.1) | 99.3 (90.5)

17. Secondary Outcome: Percentage of Participants With Other Skin Lesions of Any Grade During the First 4 Months of Treatment
Description: Other skin lesions included presence or absence of xerosis and paronychia.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 39.7 | 42.5

18. Secondary Outcome: Percentage of Participants With Other Skin Lesions During the First 4 Months of Treatment By Type
Description: Other skin lesions included xerosis and paronychia.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants
  Xerosis | 37.0 | 41.1
  Paronychia | 6.8 | 8.2

19. Secondary Outcome: Percentage of Participants With Other Skin Lesions During the First 4 Months of Treatment By Maximal Intensity
Description: Other skin lesions included xerosis and paronychia. Intensity was classified according to CTCAE grading. Grade 1=Macular or papular eruption or erythema without associated symptoms; Grade 2=Macular or papular eruption or erythema with pruritus or other associated symptoms; localized desquamation or other lesions covering <50% of BSA; Grade 3=Severe, generalized erythroderma or macular, papular, or vesicular eruption; desquamation; Grade 4=Generalized exfoliative, ulcerative, or bullous dermatitis. If a participant had several skin lesions, the maximal intensity was taken into account.
Time Frame: Days 0, 14, 28 and Months 2, 3, and 4
Population: ITT population; only participants with an adverse event classified as other skin lesion during the first 4 months were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 29 | 31
percentage of participants
  Grade 1 | 69.0 | 29.0
  Grade 2 | 24.1 | 51.6
  Grade 3 | 6.9 | 16.1
  Grade 4 | 0 | 3.2
Statistical Analysis 1: Comparison: Erlotinib + Doxycycline vs Erlotinib; Erlotinib + doxycycline vs Erlotinib: Grade 3; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel

20. Secondary Outcome: Percentage of Participants With Erlotinib Dose Reduction by Reason for Reduction
Description: Erlotinib dose adjustment was done in case of toxicity occurrence. Keratitis, diarrhea, interstitial lung disease, and other toxic occurrences determined erlotinib dose reduction. If erlotinib was previously discontinued for skin rash or diarrhea of Grade 2 and if these symptoms of Grade 2 recurred OR if the symptoms were intolerable for the participants, erlotinib was discontinued until recovery/Grade 1 then the dose was reduced of one level of 50 mg.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT population; only participants that discontinued or interrupted erlotinib were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 23 | 32
percentage of participants
  Adverse event | 80.0 | 85.7
  Investigator's decision | 0 | 2.4
  Other | 20.0 | 11.9

21. Secondary Outcome: Percentage of Participants With Doxycycline Dose Reduction by Reason for Reduction
Description: Occurrence of folliculitis-type skin rash of Grade greater than or equal to (≥)2 led to dose modification. Continuation of treatment with doxycycline after occurrence of folliculitis-type skin rash of Grade ≥2 was upon the investigator's opinion.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT population; only participants that discontinued or interrupted doxycycline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 8 | 0
percentage of participants
  Adverse event | 50.0 |
  Other | 50.0 |

22. Secondary Outcome: Percentage of Participants With Global Disease Control by Visit
Description: Disease control was determined according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria for evaluation and was defined as participants with either complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: Months 2, 4, 7, 10, and 12
Population: ITT population; number (n) = number of participants analyzed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 34 | 33
percentage of participants
  Month 2 (n=34,33) | 88.2 | 93.9
  Month 4 (n=19,25) | 89.5 | 80.0
  Month 7 (n=11,17) | 72.7 | 76.5
  Month 10 (n=7,12) | 100.0 | 66.7
  Month 12 (n=7,10) | 71.4 | 40.0

23. Secondary Outcome: Percentage of Participants by Best Global Response Under Treatment
Description: Response was determined according to the RECIST criteria for evaluation and was defined as participants with either CR, PR, SD, or progression. No CR was reported.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 58 | 58
percentage of participants
  PR | 15.5 | 10.3
  SD | 36.2 | 48.3
  Progression | 48.3 | 41.4

24. Secondary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined by the time between first intake of treatment with erlotinib and disease progression or death for any cause; estimated using Kaplan-Meier method.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 91.8 | 87.8

25. Secondary Outcome: Progression-Free Survival (PFS) - Time to Event
Description: as for outcome 24
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
days | 63.0 [56.0 to 107.0] | 70.0 [56.0 to 107.0]

26. Secondary Outcome: Percentage of Participants Estimated to be Progression Free at 4 and 12 Months
Time Frame: Months 4 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants
  4 Months | 30.1 | 31.0
  12 Months | 6.3 | 10.8

27. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined by the time between first intake of treatment with erlotinib and death for any cause; analyzed using Kaplan-Meier method.
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants | 71.2 | 67.6

28. Secondary Outcome: Overall Survival (OS) - Time to Event
Description: as for outcome 27
Time Frame: Days 0, 14, 28 and Months 2, 3, 4, 7, 10, and 12
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
days | 227.0 [153.0 to 282.0] | 251.0 [152.0 to 336.0]

29. Secondary Outcome: Percentage of Participants Estimated to be Alive at 4 and 12 Months
Time Frame: Months 4 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 73 | 74
percentage of participants
  4 Months | 68.5 | 69.7
  12 Months | 27.1 | 33.5

30. Secondary Outcome: Dermatology Life Quality Index (DLQI) Global Score
Description: Quality of life was assessed by participant's responses to a DLQI questionnaire. The DLQI is a 10-item questionnaire assessing quality of life; questions were assessed on a 4-point scale (0=not at all; 1=a little; 2=a lot; and 3=very much). The DLQI was calculated by summing the score of each question resulting in a maximum of 30 (extremely large effect on participant's life) and a minimum of 0 (no effect at all on participant's life). The higher the score, the more quality of life is impaired. Analysis was performed by visit well as at the last available value after baseline (Endpoint); change from baseline to endpoint was also determined.
Time Frame: Baseline, Days 14 and 28 and Months 2, 3, and 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 67 | 69
units on a scale
  Baseline (n=67,69) | 0.2 (0.5) | 0.2 (0.6)
  Day 14 (n=63,62) | 1.7 (3.2) | 3.7 (4.3)
  Day 28 (n=60,56) | 1.7 (2.5) | 3.4 (4.0)
  Month 2 (n=35,37) | 2.3 (4.1) | 4.3 (5.3)
  Month 3 (n=29,27) | 1.7 (2.7) | 3.2 (3.7)
  Month 4 (n=19,24) | 1.6 (3.0) | 2.6 (3.5)
  Endpoint (n=65,63) | 2.0 (3.3) | 3.4 (4.8)
  Change at Endpoint (n=35,37) | 1.9 (3.3) | 3.2 (4.8)

31. Secondary Outcome: Percentage of Participants by DLQI Global Score Classification of Disease Effect on Quality of Life
Description: Quality of life was assessed by participant's responses to a DLQI questionnaire. The DLQI is a 10-item questionnaire assessing quality of life; questions were assessed on a 4-point scale (0=not at all; 1=a little; 2=a lot; and 3=very much). The DLQI was calculated by summing the score of each question resulting in a maximum of 30 (extremely large effect on participant's life) and a minimum of 0 (no effect at all on participant's life). The higher the score, the more quality of life is impaired. The DLQI global score was classified into 5 levels: 0-1 (no effect at all), 2-5 (small effect), 6-10 (moderate effect), 11-20 (very large effect) and 21-30 (extremely large effect).
Time Frame: Baseline, Days 14 and 28 and Months 2, 3, and 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 67 | 69
percentage of participants
  Baseline, no effect (n=67,69) | 98.5 (0.5) | 97.1 (0.6)
  Baseline, small effect (n=67,69) | 1.5 (3.2) | 2.9 (4.3)
  Day 14, no effect (n=63,62) | 69.8 (2.5) | 41.9 (4.0)
  Day 14, small effect (n=63,62) | 27.0 (3.3) | 30.6 (4.8)
  Day 14, moderate effect (n=63,62) | 0.0 (4.1) | 21.0 (5.3)
  Day 14, very large effect (n=63,62) | 1.6 (2.7) | 6.5 (3.7)
  Day 14, extremely large effect (n=63,62) | 1.6 (3.0) | 0.0 (3.5)
  Day 28, no effect (n=60,56) | 66.7 | 41.1
  Day 28, small effect (n=60,56) | 25.0 | 35.7
  Day 28, moderate effect (n=60,56) | 8.3 | 19.6
  Day 28, very large effect (n=60,56) | 0.0 | 1.8
  Day 28, extremely large effect (n=60,56) | 0.0 | 1.8
  Month 2, no effect (n=35,37) | 65.7 | 40.5
  Month 2, small effect (n=35,37) | 22.9 | 27.0
  Month 2, moderate effect (n=35,37) | 5.7 | 21.6
  Month 2, very large effect (n=35,37) | 5.7 | 8.1
  Month 2, extremely large effect (n=35,37) | 0.0 | 2.7
  Month 3, no effect (n=29,27) | 69.0 | 37.0
  Month 3, small effect (n=29,27) | 27.6 | 44.4
  Month 3, moderate effect (n=29,27) | 0.0 | 11.1
  Month 3, very large effect (n=29,27) | 3.4 | 7.4
  Month 4, no effect (n=19,24) | 78.9 | 50.0
  Month 4, small effect (n=19,24) | 15.8 | 41.7
  Month 4, very large effect (n=19,24) | 5.3 | 8.3

32. Secondary Outcome: Quality of Life Score as Assessed by Visual Analog Scale (VAS)
Description: Quality of life was assessed by participant's responses to a VAS questionnaire - (evaluation of satisfaction with skin status). VAS was measured on a 100 millimeter (mm) scale where 0 = not at all satisfied and 100 = very satisfied. Participants were asked to mark the line corresponding to their satisfaction at each visit and the distance from the left edge was measured. A negative change from baseline indicates improvement. Analysis was performed by visit well as at the last available value after baseline (Endpoint).
Time Frame: Baseline, Days 14 and 28, and Months 2, 3, and 4
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Number analyzed (Participants) | 64 | 68
mm
  Baseline (n=64,68) | 81.4 (23.7) | 87.8 (19.6)
  Day 14 (n=62,63) | 68.8 (26.6) | 51.0 (34.5)
  Change at Day 14 (n=59,61) | -16.2 (28.5) | -39.2 (37.8)
  Day 28 (n=59,56) | 66.5 (27.2) | 54.8 (27.0)
  Change at Day 28 (n=55,54) | -15.5 (28.8) | -35.1 (27.8)
  Month 2 (n=36,36) | 68.9 (22.8) | 52.6 (27.4)
  Month 3 (n=28,27) | 63.5 (21.4) | 56.1 (31.7)
  Month 4 (n=18,24) | 71.8 (20.9) | 59.9 (29.7)
  Endpoint (n=65,64) | 64.0 (26.6) | 58.3 (30.8)
  Change at Endpoint (n=60,62) | -18.1 (27.7) | -30.4 (31.4)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded continuously until 30 days after the last treatment administration.
Arm/Group | Erlotinib + Doxycycline | Erlotinib
Serious Adverse Events (participants affected / at risk) | 18/73 | 24/74
Other Adverse Events (participants affected / at risk) | 71/73 | 69/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Doxycycline (N=73) | Erlotinib (N=74)
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
General physical health deterioration (General disorders) | 4 | 6
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Chest pain (General disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Xerosis (General disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Headache (Nervous system disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Doxycycline (N=73) | Erlotinib (N=74)
Folliculitis (Skin and subcutaneous tissue disorders) | 53 | 58
Paronychia (Skin and subcutaneous tissue disorders) | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 26 | 34
Vomiting (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 8 | 8
Constipation (Gastrointestinal disorders) | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Stomatitis (Gastrointestinal disorders) | 8 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Xerosis (General disorders) | 28 | 30
Asthenia (General disorders) | 5 | 9
General physical health deterioration (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 3 | 1
Chest pain (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Catheter site inflammation (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Fungal skin infection (Infections and infestations) | 2 | 2
Oral fungal infection (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 6
Dry eye (Eye disorders) | 2 | 1
Eye pruritus (Eye disorders) | 1 | 1
Growth of eyelashes (Eye disorders) | 0 | 2
Eye irritation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Visual distrubance (Eye disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Sciatica (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Aphonia (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Epiduritis (Nervous system disorders) | 1 | 0
Facial neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 4
Blood bilirubin increased (Investigations) | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Periphlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 3
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.